CLINICAL TRIAL: NCT03192605
Title: The Effect of Wild Blueberry Consumption on Diabetes: Evaluation of Glucose Regulation, Gastrointestinal Hormones and Satiety in Healthy Adults
Brief Title: The Effect of Wild Blueberry Consumption on Glucose Regulation in Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Prince Edward Island (Other)
Responsible Party: Principal Investigator, Kim Stote, Research Chair of Nutrisciences and Health, University of Prince Edward Island
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: UPEI
Record Dates: First submitted 2017-06-16; First posted 2017-06-20 (Actual); Last update posted 2017-06-20 (Actual); Status verified 2017-06

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — blueberry extract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Blueberry (Experimental): 150 grams wild blueberries
  Interventions: Other: Blueberry
- Placebo (Placebo Comparator): Placebo control
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Blueberry — Blueberry - 150 grams wild blueberries (whole fruit)
  Arms: Blueberry
Other: Placebo — Placebo - matched for calories and fiber
  Arms: Placebo

SUMMARY:
The objective of the study is to determine how wild blueberry consumption affects glucose regulation, gastrointestinal hormones and satiety in healthy adults.

DETAILED DESCRIPTION:
Healthy men and women (ages 21 - 65 years) were recruited to take part in a randomized, placebo controlled crossover design study. Subjects were screened to determine their health status (e.g. height, weight, body mass index, blood pressure and medical history). Subjects were randomly assigned to a sequence of two treatments with two study periods. The treatments are frozen wild blueberries and a placebo developed to match calories and fiber of the frozen wild blueberries. The subjects were asked to avoid high polyphenol foods in their typical diet for 7 days and consume one of the two treatments as a dietary intervention. After the seventh day subjects consumed a test meal along with either the wild blueberry or placebo. Blood was collected to determine glucose and satiety hormone levels.

ELIGIBILITY:
Inclusion Criteria:

* Male or female

Exclusion Criteria:

* BMI < 20 and > 30 kg/m²
* Pregnant women or women who plan on becoming pregnant during the study
* Postpartum women
* Lactating women
* Diabetes Mellitus
* Kidney disease
* Liver disease
* GI Disease
* Certain cancers
* Smokers
* Blueberry allergies

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2017-06-02 (Actual); Study Completion 2017-06-02 (Actual)

PRIMARY OUTCOMES:
Glucose (mmol/L) | Change from baseline 0 hours and 2 hours
  Plasma glucose

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Gottschall-Pass, PhD, Principal Investigator — University of Prince Edward Island
Locations (1):
- University of Prince Edward Island, Health Sciences, Charlottetown, Prince Edward Island, Canada

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared as requested by other researchers. It may be made available by June 2018.